CLINICAL TRIAL: NCT05781321
Title: Stereotactic Accelerated Radiotherapy in GlioblastomA (SAGA)
Brief Title: Short Course Radiotherapy for the Treatment of Patients With Glioblastoma, SAGA Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GMROR2261; NCI-2023-01559 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GMROR2261 (Other: Mayo Clinic Radiation Oncology); 22-006990 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2023-02-27; First posted 2023-03-23 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — fluorodopa F 18; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation; Temozolomide; Specimen Handling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The MRI scan indicating progressive disease will be fused with our treatment planning scan and the region of progression will be contoured by an investigator blinded to the GTV_MRI, T2_FLAIR_NCET, GTV_PET, PTV_high, and isodose lines.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (short course RT) (Experimental): Patients undergo short course RT for 5-10 fractions over 1-2 weeks on study. Patients also receive temozolomide PO on days 1-5 every 28 days during radiation therapy. Starting one month post-radiation, patients continue temozolomide on days 1-5 every 28 days for up to 5 adjuvant cycles in the absence of disease progression or unacceptable toxicity. Patients undergo PET/CT with 18-F-DOPA administered IV prior to RT on study, and undergo MRI prior to RT and throughout the trial. Patients may optionally undergo blood sample collection during screening and on the trial.
  Interventions: Radiation: Accelerated Hypofractionated Radiation Therapy; Procedure: Computed Tomography; Drug: Fluorodopa F 18; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Temozolomide; Procedure: Biospecimen Collection
- Arm B (standard course RT) (Active Comparator): Patients undergo standard course RT for 15-30 fractions over 3-6 weeks on study. Patients also receive temozolomide PO QD concurrently with radiation therapy and for up to 6 adjuvant cycles in the absence of disease progression or unacceptable toxicity. Patients undergo PET/CT with 18-F-DOPA administered IV prior to RT on study, and undergo MRI prior to RT and throughout the trial. Patients may optionally undergo blood sample collection during screening and on the trial.
  Interventions: Procedure: Computed Tomography; Drug: Fluorodopa F 18; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy; Drug: Temozolomide; Procedure: Biospecimen Collection

INTERVENTIONS:
Radiation: Accelerated Hypofractionated Radiation Therapy — Undergo short course RT
  Other Names: AHF-RT; AHRT
  Arms: Arm A (short course RT)
Procedure: Computed Tomography — Undergo CT simulation
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Drug: Fluorodopa F 18 — Given IV
  Other Names: (18F)FDOPA; 18F-DOPA; 18F-FDOPA; 3-(2-Fluoro-(sup 18)F-4,5-dihydroxyphenyl)-L-alanine; 6-(18F)Fluoro-L-DOPA; Fluorine F 18 Fluorodopa; Fluorine-18-fluoro-L-DOPA; Fluorodopa (18F); FLUORODOPA F-18; L-6-(18F)Fluoro-DOPA
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Quality-of-Life Assessment — Ancillary studies
Other: Questionnaire Administration — Complete questionnaires
Radiation: Radiation Therapy — Undergo standard course RT
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Arm B (standard course RT)
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection

SUMMARY:
This phase II trial compares the effect of short course radiotherapy (RT) to standard course RT for the treatment of patients diagnosed with glioblastoma (GBM). The researchers want to learn whether the shorter course treatment is non-inferior (not worse than the standard of care), for patients with GBM. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors. Short course radiotherapy delivers higher doses of radiation over a shorter period of time and may kill more tumor cells and have fewer side effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To demonstrate non-inferior 12-month overall survival (OS) of patients with GBM treated with dose escalated hypofractionated radiotherapy compared to standard of care.

SECONDARY OBJECTIVES:

I. To demonstrate the safety of short-course radiotherapy via physician-reported grade (G) 3+ toxicity.

II. To explore patient-reported outcomes to demonstrate favorable quality of life with short-course radiotherapy for GBM.

III. To analyze the impact of shortening the treatment duration on treatment related lymphopenia and absolute lymphocyte counts.

EXPLORATORY OBJECTIVES:

I. To determine the cost-effectiveness of the 5-fraction treatment regimen compared to standard of care.

II. To explore the impact on the immune system with the 5-fraction treatment regimen. Immune phenotyping will be assessed by Flow Cytometry and cytometry by flight (CyTOF).

III. To analyze series of cytokine levels over time. IV. To assess patterns of failure, specifically focusing on differences in volume delineation via Fluorodopa F 18 (FDOPA) and magnetic resonance imaging (MRI) and recurrences in-field versus (vs.) out of field.

V. To conduct a subgroup analysis for just patients =< 65 cc. VI. To conduct a subgroup analysis for just patients with and without tumor treating fields.

VII. To analyze patient demographic data compared to historical controls to determine whether the short-course treatment regimen improves access to underserved populations.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients undergo short course RT for 5-10 fractions over 1-2 weeks on study. Patients also receive temozolomide orally (PO) on days 1-5 every 28 days during radiation therapy. Starting one month post-radiation, patients continue temozolomide on days 1-5 every 28 days for up to 5 adjuvant cycles in the absence of disease progression or unacceptable toxicity.

ARM B: Patients undergo standard course RT for 15-30 fractions over 3-6 weeks on study. Patients also receive temozolomide PO daily (QD) concurrently with radiation therapy and for up to 6 adjuvant cycles in the absence of disease progression or unacceptable toxicity.

All patients undergo positron emission tomography/computed tomography (PET/CT) with 18-F-DOPA administered intravenously (IV) prior to RT on study, and undergo MRI prior to RT and throughout the trial. Patients may optionally undergo blood sample collection during screening and on the trial.

After completion of study treatment, patients are followed up every 2 months for the first year, every 3 months for the second year, and every 4 months for the third year. After 3 years, clinical outcomes are monitored at least once a year until 5 years after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Histological and/or molecular confirmation of glioblastoma
* Eastern Oncology Group (ECOG) performance status (PS) =< 3
* Ability to complete questionnaire(s) by themselves or with assistance
* Provide written informed consent or have a legally authorized representative (LAR) who is responsible for the care and well-being of the potential study participant, provide consent
* Willing to return to enrolling institution for follow-up either in-person or by video visit
* Postoperative/post-biopsy tumor plus surgical bed size =< 6 cm in maximum diameter. This measurement includes both the enhancing region identified via T1 MRI with contrast, as well as the surgical cavity

Exclusion Criteria:

* Unable to undergo MRI scans with contrast
* Unable to undergo an 18F-DOPA-PET scan (e.g., Parkinson's Disease, taking carbidopa/levodopa and/or less than 48 hours from discontinuance)
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Tumors with IDH mutation
* Previous brain radiation therapy
* Patients who will not receive any radiation treatment or who will receive radiation treatment elsewhere (Note: radiotherapy can be given on the trial at Mayo Clinic facilities in Rochester, Arizona, or Florida, as well as at the Mayo Clinic Health System sites). Temozolomide, however, can be provided by another institution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2026-07-02 (Estimated); Study Completion 2028-07-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients alive [overall survival (OS)] at 12 months | Up to 12 months after enrollment
  OS is defined as the time from study registration to death due to any cause.

SECONDARY OUTCOMES:
Proportion of patients whose radiation oncologist reported a grade 3+ toxicity | 30-, 90-, and 180-days post-radiotherapy (RT)
  Pretreatment symptoms/conditions will be graded at enrollment by the radiation oncology team and updated at each evaluation. Adverse Events will be calculated using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Quality of life: EORTC QLQ-C30 | From baseline up to 3 years
  Assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30), a 30 item questionnaire used to assess quality of life in cancer patients. Questions are answered using a 4-point Likert scale where 1=not at all and 4=very much, except for two items which use a 7-point scale where 1=very poor and 7=excellent. Higher scores on the questions answered 1-4 indicate more severe symptoms and greater difficulty. Higher scores on the 1-7 scales indicate better overall health and quality of life.
Quality of life: EORTC QLQ-BN20 | From baseline up to 3 years
  Assessed using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Brain Neoplasm (QLQ-BN20), which consists of 20 questions answered using a 4-point Likert scale where 1=not at all and 4=very much. Higher scores reflect more severe symptoms.
Lymphocyte count | From baseline up to 3 years
  Assessed by blood test, lymphocyte count will be compared between arms by change in count from pretreatment to end of RT.

CONTACTS AND LOCATIONS:
Overall Officials: William G. Breen, MD, Principal Investigator — Mayo Clinic in Rochester; Roman O. Kowalchuk, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (8):
- United States (8):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Mayo Clinic Radiation Therapy - Northfield, Northfield, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mayo Clinic Health System-Eau Claire, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials